CLINICAL TRIAL: NCT02891460
Title: Evaluation of the Clinical Response of Mitomycin-C (MMC) Embedded in Hydrogel (TC-3) in Comparison to Mitomycin C in Saline, When Administered Intravesically, Pre-TURBT in Non Muscle Invasive Bladder Cancer (NMIBC) Patients. Muscle Invasive Bladder Cancer (NMIBC) Patients
Brief Title: Pilot Study to Evaluate the Clinical Response to Mitomycin-C in Hydrogel (TC-3) Administered Intravesically in NMIBC Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC-3 /2012 / P2
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Urinary Bladder Neoplasms; Urologic Neoplasms; Neoplasms; Urinary Bladder Diseases; Urologic Diseases
Keywords: Mitomycin C; MMC; NMIBC; Non Muscle Invasive Bladder Cancer; Hydrogel Reverse thermal gelation; Drug retention; Urinary Bladder Neoplasms; Urologic Neoplasms; Urinary Bladder Diseases; Urologic Diseases
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urologic Neoplasms; Neoplasms; Urinary Bladder Diseases; Urologic Diseases; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 40 mg MMC in 40 mL TC-3. (Experimental): TC-3 gel mixed with Mitomycin C (MMC) Six weekly intravesical instillations of 40 ml of TC-3 gel mixed with 40 mg MMC will be instilled using catheter.
  Interventions: Device: 40 mg MMC in 40 mL TC-3.
- 80 mg MMC in 40 mL TC-3. (Experimental): TC-3 gel mixed with Mitomycin C (MMC) Six weekly intravesical instillations of 40 ml of TC-3 gel mixed with 80 mg MMC will be instilled using catheter.
  Interventions: Device: 80 mg MMC in 40 mL TC-3.

INTERVENTIONS:
Device: 40 mg MMC in 40 mL TC-3. — A reverse thermal biodegradable gel (TC-3) (low viscosity at 5°C gel appearance at body temperature) for drug retention in the urinary bladder.
  Other Names: MMC-Gel
  Arms: 40 mg MMC in 40 mL TC-3.
Device: 80 mg MMC in 40 mL TC-3. — A reverse thermal biodegradable gel (TC-3) (low viscosity at 5°C gel appearance at body temperature) for drug retention in the urinary bladder.
  Other Names: MMC-Gel
  Arms: 80 mg MMC in 40 mL TC-3.

SUMMARY:
The purpose of this study is to evaluate the clinical response of the tumors within the bladder of recurrent NMIBC patients to Mitomycin-C embedded in UroGen Pharma's (known at that time as TheraCoat Ltd.) TC-3 Sterile Hydrogel (TC-3) and to evaluate the patency of ureters 6 hr post instillation.

DETAILED DESCRIPTION:
An open label, successive dose escalation trial in subjects with Non Muscle Invasive Bladder Cancer (NMIBC), designed to evaluate the clinical response of low-intermediate risk tumors within the bladder to Mitomycin-C embedded in TC-3 Sterile Hydrogel (TC-3), administered intravesically, prior to TURBT in NMIBC subjects.

Eligible subjects with NMIBC will be recruited to the trial following the initial diagnostic cystoscopy. During the diagnostic cystoscopy, the number of tumor lesions, their size and location will be documented and recorded with video or photo cystoscopy.

A baseline cystoscopy will be conducted in all subjects for the evaluation of number of tumors and their diameters, and for mapping of their location. Baseline blood samples for liver and renal functions, as well as for complete blood count (CBC) and coagulation tests will be drawn prior to instillation to ensure eligibility and to serve as a reference point for systemic safety follow-up.

A future TURBT has been planned for 8-10 weeks post screening. Enrolled subjects will be treated successively with 40mg MMC in 40 mL TC-3 (the first 6 subjects) and with 80 mg MMC in 40 mL TC-3 (the following 12 subjects). At treatment session initiation, an 18-20 Fr two-way catheter will be inserted into the subject's bladder in order to completely empty the bladder of urine. Thereafter, a volume of 40 mL of cooled TC-3 mixed with 40 mg or 80 mg of MMC will be instilled through the catheter into the bladder of the subject. The catheter will then be ligated for twenty minutes, after which it will be drawn out of the bladder and the subject was will be allowed to urinate freely.

The subjects will undergo six weekly bladder instillations according to their assigned treatment of either 40 mg MMC (Group A) or 80 mg MMC (Group B) in 40 mL of TC-3. Following completion of instillation treatment series, there will be a 2-4 weeks healing period prior to next follow up visit (overall 10-12 weeks post screening). During 2-4 weeks follow-up (FU) visit, the lesions' status will be examined under cystoscopy. For subjects who will appear to have complete response (CR), this will be confirmed based on histological results. For subjects that will not be classified as having CR, decision about performance of TURBT or giving additional treatment will be at the PI's discretion.

Following 2-4 week FU visit, subjects will be managed according to their local standard guidelines. All patients will attempt to be followed up for 12 months following 2-4 weeks FU within the trial. These visits will be documented and data regarding recurrence and progression will be collected. Moreover, biopsy slides prior (when available), and following treatment will be collected and analyzed by an independent uro-pathologist.

ELIGIBILITY:
Main Inclusion criteria:

1. Single or multiple tumors (n≤7)
2. Recurrent or Naive tumor.
3. No prior history of T1 and/or Tis
4. At least one tumor >1mm.
5. Largest tumor diameter ≤ 30mm
6. Cystoscopic appearance of papillary Low or high grade tumor

Main Exclusion Criteria:

1. Carcinoma In Situ (CIS)
2. Over 7 lesions
3. Lesion is larger than 30mm in diameter
4. Cystoscopic appearance suspicious for Tis
5. Tumor located in prostatic urethra
6. Previous systemic chemotherapy or pelvic radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Subject's degree of response at 2-4 weeks post-treatment | 9-11 weeks
  Cystoscopic and pathological effect of pre-TURBT intravesical instillations with 40 or 80 mg of MMC mixed with 40cc TC-3 Hydrogel on bladder lesion(s) of NMIBC patients
Adverse events (AE) including serious adverse events (SAE) | 1.2 years
Anesthesia information | 7 weeks
  Information of whether anesthesia was used during the treatment will be collected
Blood and urine tests | 9-11 weeks
  Blood and urine tests (including urine culture test) be be collected
The degree of pain during treatment | 7 weeks
  The degree of pain subject felt at the time the drug will be injected to the bladder will be collected (VAS)
Gel clearance and urinary patency | 7 weeks
  Data regarding gel clearance and adverse urinary patency post instillation will be obtained based on the "post instillation telephone follow-up" set of questions.

SECONDARY OUTCOMES:
Tumor recurrence rate during 12 months post- 2-4 week follow-up visit in complete response (CR) subjects. | 1.2 years
Lesion Mass by time point (Screening and 2-4 weeks post-treatment) | 9-11 weeks
  Lesion mass will consider the number and size of the papillary lesion, and will be described at Screening and in 2-4 weeks follow-up visit

OTHER OUTCOMES:
Subjects' satisfaction with the treatment | 9-11 weeks
  Subjects' satisfaction with the treatment will be measured using an 8-item satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sudhir Rawal, MD, Principal Investigator — Rajiv Gandhi Cancer Institute & Research Center
Locations (1):
- Rajiv Gandhi Cancer Institute & Research Center, Delhi, New Delhi, India

REFERENCES:
- See also: UroGen pharma official website — http://www.urogen.com/